CLINICAL TRIAL: NCT04419376
Title: Driving Pressure and Mortality: in the Pediatric Intensive Care Unit (PICU)
Status: Completed | Type: Observational
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Ekin soydan, Principal Investigator, Dr. Behcet Uz Children's Hospital
Other Study IDs: 2019-344
Record Dates: First submitted 2020-06-01; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: ARDS, Human; Respiratory Failure
Keywords: Driving pressure; mortality; Pediatric intensive care unit; Pediatric acute respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — All patients were ventilated with volume control (VCV) or pressure control (PCV) mode during the hospitalization. İn order to measure the driving pressure of patients, Pplat was measured in the mechanical ventilator every 12 hours using an inspiratory hold maneuver. The average Pplat was calculated using the mean of 2 measurements within 24 hours. Then, the total PEEP was measured by expiratory hold maneuver and ΔP was calculated with the Pplat-PEEP formula.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pARDS: Within 7 days of known clinical insult Respiratory failure not fully explained by cardiac failure or fluid overload chest imaging findings of new infiltrate(s) consistent with acute pulmonary parenchymal disease patients with an oxygenation index (OI) ([FIO2 × mean airway pressure × 100]/PaO2) above 4
  Interventions: Device: driving pressure
- Patients with non-pARDS: non-pARDS patients who received mechanical ventilation support due to respiratory failure.
  Interventions: Device: driving pressure

INTERVENTIONS:
Device: driving pressure — Mechanically ventilated patients (via ETT or trachestomy) were recorded for patients whose ventilation duration lasted at least 24 hours.We divided the patients into two groups by calculating the oxygenation index (OI): [mean airway pressure(MAP) × fraction of inspired oxygen (FiO2) ]/ partial pressure of oxygen in arterial blood (PaO2) × 100) used in the classification of PALICC, including pARDS and non-pARDS.

SUMMARY:
Respiratory failure is one of the most common causes of both hospitalization and mortality in patients in the pediatric intensive care unit (PICU). Recently, it is recommended to target driving pressure (ΔP) in patients with ARDS to achieve better results with the administration of optimal mechanical ventilation. In many studies, higher ΔP was associated with mortality in adult ARDS patients; non-ARDS patients' studies showing the relationship between driving pressure and mortality are few, but contradictory results have come out.

This study aimed to determine whether ΔP was associated with mortality in pediatric patients diagnosed as pARDS and non-pARDS who received mechanical ventilation support due to respiratory failure. Patients who received invasive mechanical ventilation support due to respiratory failure in the pediatric intensive care unit over 1 month and under 18 years were included in our study Driving pressure was significantly associated with an increased risk of mortality among mechanically ventilated both pARDS and non-pARDS patients. Future prospective randomized clinical trials are needed to determine a protocol targeting DP can be developed and defining optimum cutoff values.

DETAILED DESCRIPTION:
Respiratory failure is one of the most common causes of both hospitalization and mortality in patients in the pediatric intensive care unit (PICU). Recently, it is recommended to target driving pressure (ΔP) in patients with ARDS to achieve better results with the administration of optimal mechanical ventilation. ΔP is calculated as the difference between Plateau pressure (Pplat) and positive end-expiratory pressure (PEEP) and is determined by the ratio of the tidal volume to the compliance of the respiratory system (ΔP = Pplat - PEEP = VT/CRS). ΔP estimates how much mechanical strain (dynamic strain) the tidal volume causes in the lung. It is a non-invasive and simple method and can be easily calculated at the bedside. In many studies, higher ΔP was associated with mortality in adult ARDS patients; non-ARDS patients' studies showing the relationship between driving pressure and mortality are few, but contradictory results have come out.

This study aimed to determine whether ΔP was associated with mortality in pediatric patients diagnosed as pARDS and non-pARDS who received mechanical ventilation support due to respiratory failure.

Single-center, prospective, observational study of patients admitted to pediatric intensive care units (PICU) in Turkey. In our study, the ethics committee was approved by The Health Sciences University Izmir Behcet Uz Child Health and Diseases education and research hospital ethics committee (protocol no: 2019-344).In our study, patients who received invasive mechanical ventilation support due to respiratory failure in the pediatric intensive care unit over 1 month and under 18 years were included in the study between March 2018 and April 2020. Mechanically ventilated patients (via ETT or trachestomy) were recorded for patients whose ventilation duration lasted at least 24 hours. We divided the patients into two groups by calculating the oxygenation index (OI): [mean airway pressure(MAP) × fraction of inspired oxygen (FiO2) ]/ partial pressure of oxygen in arterial blood (PaO2) × 100) used in the classification of PALICC, including ARDS and non-ARDS. PARDS definition was also identified based on the PALICC criteria. Data were prospectively recorded on day 1 including patient demographics, ventilator settings (VT, VT / ideal body weight (IBW), respiratory rate (RR), peak inspiratory pressure (PIP), plateau pressure (Pplat), mean airway pressure (Pmean), minute volume (VE), end-expiratory pressure (PEEP), static compliance (Cstat), fraction of inspired oxygen FIO2, inspiratory time ( IT), expiratory time (ET) and we calculated oxygenation index (OI), cstat (VT/∆P), partial pressure of oxygen in arterial blood (PaO2) /FiO2, driving pressure (ΔP), the pediatric index of mortality (PRISM) III scores and pediatric sequential organ failure assessment (pSOFA) scores.

All patients were ventilated with volume control (VCV) or pressure control (PCV) mode during the hospitalization. İn order to measure the driving pressure of patients, Pplat was measured in the mechanical ventilator every 12 hours using an inspiratory hold maneuver. The average Pplat was calculated using the mean of 2 measurements within 24 hours. Then, the total PEEP was measured by expiratory hold maneuver and ΔP was calculated with the Pplat-PEEP formula. Patients were followed for 30 days until hospital discharge. We used ΔP compared to other mechanic ventilator parameters between survivors and non-survivors at day 30. Besides, ΔP and other parameters of patients in the ARDS and non-ARDS groups were compared with their 30-day mortality.

Statistical Analyses Primarily, we evaluated the relationship between ΔP and mortality in patients with ARDS and non-ARDS. Our second target was to evaluate the relationship between mortality and ΔP and other mechanical ventilator parameters.

Driving pressure and other lung dynamics; according to the type and distribution of the data was compared with chi-square, Wilcoxon, Independent-T-test or Mann-Whitney-U test and p <0.05 was considered statistically significant. The strength of the association between the two variables was measured using the correlation coefficient. We used Pearson correlation to parametric variable and Spearman correlation to the nonparametric variable to detect covariances before logistic regression analysis. We evaluated with spearman's correlation analysis to detect covariances before logistic regression analysis. Parameters found significant with mortality in univariate analyzes were evaluated by Logistic Regression analysis. (odds ratio [OR] and 95 % confidence intervals [CI]) Model fit was assessed using Hosmer-Lemeshow statistics.

For the multivariable analysis, we identified covariates that may be associated with mortality. VT /IBW, PaO2, OI, FiO2, PRISM III score, Days of ventilation and pSOFA score were not collinear with ΔP. We did not include Pplat, PIP, Pmean in logistic regression models containing ΔP given concerns for collinearity Individual covariates included age, gender, PRISM III score, PaO2, OI, FiO2, Days of ventilation and pSOFA score. We created 3 other modeling analyzes for Pplat, PIP, Pmean, because of collinearity with driving pressure. We evaluated this model to determine the best parameter related to mortality in whole patients under mechanical ventilation support due to respiratory failure. ΔP cut off (13 cmH2O) values in adult studies in the literature were categorized and mortality was estimated by a receiver operating characteristic (ROC). We performed all statistical analyses using IBM SPSS Statistics for Windows version 22 (Armonk, NY) for analysis.

Mechanical ventilation is one of the most common indications for admission to a pediatric intensive care unit (PICU), with up to 64% of admitted children requiring mechanical ventilation. Driving pressure (ΔP), which is calculated as end-inspiratory plateau pressure (Pplat) minus applied positive end-expiratory pressure (PEEP) and is equivalent to the ratio between the VT and compliance of the respiratory system, can reduce mortality with children who received mechanical ventilator support due to respiratory failure. ΔP is a non-invasive and simple method and can be easily calculated at the bedside.

Recent data in the adult ARDS population have shown that the ΔP is most related to mortality. Our study, we have shown that the ΔP on day 1 was associated with hospital mortality in with pARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* In our study, patients who received invasive mechanical ventilation support for at least 24 hours due to respiratory failure in the pediatric intensive care unit over 1 month and under 18 years were included in the study between March 2018 and April 2020.

Exclusion Criteria:

* patients who died within the first 24 hours and patients whose desired respiratory mechanics were not measured and data deficiencies were detected

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: In our study, patients who received invasive mechanical ventilation support due to respiratory failure in the pediatric intensive care unit over 1 month and under 18 years were included in the study between March 2018 and April 2020.
  Mechanically ventilated patients (via ETT or trachestomy) were recorded for patients whose ventilation duration lasted at least 24 hours. We divided the patients into two groups by calculating the oxygenation index (OI): [mean airway pressure(MAP) × fraction of inspired oxygen (FiO2) ]/ partial pressure of oxygen in arterial blood (PaO2) × 100) used in the classification of PALICC, including ARDS and non-ARDS.
Sampling Method: Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
Driving pressure and mortality with all patients | march 2018-april 2020
  Driving pressure and other lung dynamics; according to the type and distribution of the data was compared with chi-square, Wilcoxon, Independent-T-test or Mann-Whitney-U test and p <0.05 was considered statistically significant.

SECONDARY OUTCOMES:
Driving pressure with mortality in patients with pARDS and non-pARDS patients | march 2018-april 2020
  we conducted separately to determine the relationship between ΔP and mortality in patients non-ARDS and ARDS

CONTACTS AND LOCATIONS:
Overall Officials: ekin soydan, Principal Investigator — Investigator
Locations (1):
- The Health Sciences University Izmir Behçet Uz Child Health and Diseases education and research hospital, Izmir, Turkey/izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
we will share our data in the future

REFERENCES:
- [Result] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Result] Santschi M, Jouvet P, Leclerc F, Gauvin F, Newth CJ, Carroll CL, Flori H, Tasker RC, Rimensberger PC, Randolph AG; PALIVE Investigators; Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI); European Society of Pediatric and Neonatal Intensive Care (ESPNIC). Acute lung injury in children: therapeutic practice and feasibility of international clinical trials. Pediatr Crit Care Med. 2010 Nov;11(6):681-9. doi: 10.1097/PCC.0b013e3181d904c0. PMID 20228688
- [Result] Pediatric Acute Lung Injury Consensus Conference Group. Pediatric acute respiratory distress syndrome: consensus recommendations from the Pediatric Acute Lung Injury Consensus Conference. Pediatr Crit Care Med. 2015 Jun;16(5):428-39. doi: 10.1097/PCC.0000000000000350. PMID 25647235
- [Result] Kneyber MCJ, de Luca D, Calderini E, Jarreau PH, Javouhey E, Lopez-Herce J, Hammer J, Macrae D, Markhorst DG, Medina A, Pons-Odena M, Racca F, Wolf G, Biban P, Brierley J, Rimensberger PC; section Respiratory Failure of the European Society for Paediatric and Neonatal Intensive Care. Recommendations for mechanical ventilation of critically ill children from the Paediatric Mechanical Ventilation Consensus Conference (PEMVECC). Intensive Care Med. 2017 Dec;43(12):1764-1780. doi: 10.1007/s00134-017-4920-z. Epub 2017 Sep 22. PMID 28936698
- [Result] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Result] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Result] Guo L, Xie J, Huang Y, Pan C, Yang Y, Qiu H, Liu L. Higher PEEP improves outcomes in ARDS patients with clinically objective positive oxygenation response to PEEP: a systematic review and meta-analysis. BMC Anesthesiol. 2018 Nov 17;18(1):172. doi: 10.1186/s12871-018-0631-4. PMID 30447683
- [Result] Khemani RG, Conti D, Alonzo TA, Bart RD 3rd, Newth CJ. Effect of tidal volume in children with acute hypoxemic respiratory failure. Intensive Care Med. 2009 Aug;35(8):1428-37. doi: 10.1007/s00134-009-1527-z. Epub 2009 Jun 17. PMID 19533092
- [Result] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Result] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Result] Aoyama H, Pettenuzzo T, Aoyama K, Pinto R, Englesakis M, Fan E. Association of Driving Pressure With Mortality Among Ventilated Patients With Acute Respiratory Distress Syndrome: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Feb;46(2):300-306. doi: 10.1097/CCM.0000000000002838. PMID 29135500
- [Result] Chen Z, Wei X, Liu G, Tai Q, Zheng D, Xie W, Chen L, Wang G, Sun JQ, Wang S, Liu N, Lv H, Zuo L. Higher vs. Lower DP for Ventilated Patients with Acute Respiratory Distress Syndrome: A Systematic Review and Meta-Analysis. Emerg Med Int. 2019 Jul 18;2019:4654705. doi: 10.1155/2019/4654705. eCollection 2019. PMID 31396419
- [Result] Guerin C, Papazian L, Reignier J, Ayzac L, Loundou A, Forel JM; investigators of the Acurasys and Proseva trials. Effect of driving pressure on mortality in ARDS patients during lung protective mechanical ventilation in two randomized controlled trials. Crit Care. 2016 Nov 29;20(1):384. doi: 10.1186/s13054-016-1556-2. PMID 27894328
- [Result] Lanspa MJ, Peltan ID, Jacobs JR, Sorensen JS, Carpenter L, Ferraro JP, Brown SM, Berry JG, Srivastava R, Grissom CK. Driving pressure is not associated with mortality in mechanically ventilated patients without ARDS. Crit Care. 2019 Dec 27;23(1):424. doi: 10.1186/s13054-019-2698-9. PMID 31881909
- [Result] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Result] Flori HR, Glidden DV, Rutherford GW, Matthay MA. Pediatric acute lung injury: prospective evaluation of risk factors associated with mortality. Am J Respir Crit Care Med. 2005 May 1;171(9):995-1001. doi: 10.1164/rccm.200404-544OC. Epub 2004 Dec 23. PMID 15618461
- [Result] Dahlem P, van Aalderen WM, Hamaker ME, Dijkgraaf MG, Bos AP. Incidence and short-term outcome of acute lung injury in mechanically ventilated children. Eur Respir J. 2003 Dec;22(6):980-5. doi: 10.1183/09031936.03.00003303. PMID 14680089
- [Result] Schmidt MFS, Amaral ACKB, Fan E, Rubenfeld GD. Driving Pressure and Hospital Mortality in Patients Without ARDS: A Cohort Study. Chest. 2018 Jan;153(1):46-54. doi: 10.1016/j.chest.2017.10.004. Epub 2017 Oct 14. PMID 29037528
- [Result] Chiumello D, Carlesso E, Brioni M, Cressoni M. Airway driving pressure and lung stress in ARDS patients. Crit Care. 2016 Aug 22;20:276. doi: 10.1186/s13054-016-1446-7. PMID 27545828
- [Result] Raymondos K, Dirks T, Quintel M, Molitoris U, Ahrens J, Dieck T, Johanning K, Henzler D, Rossaint R, Putensen C, Wrigge H, Wittich R, Ragaller M, Bein T, Beiderlinden M, Sanmann M, Rabe C, Schlechtweg J, Holler M, Frutos-Vivar F, Esteban A, Hecker H, Rosseau S, von Dossow V, Spies C, Welte T, Piepenbrock S, Weber-Carstens S. Outcome of acute respiratory distress syndrome in university and non-university hospitals in Germany. Crit Care. 2017 May 30;21(1):122. doi: 10.1186/s13054-017-1687-0. PMID 28554331
- [Result] Farias JA, Frutos F, Esteban A, Flores JC, Retta A, Baltodano A, Alia I, Hatzis T, Olazarri F, Petros A, Johnson M. What is the daily practice of mechanical ventilation in pediatric intensive care units? A multicenter study. Intensive Care Med. 2004 May;30(5):918-25. doi: 10.1007/s00134-004-2225-5. Epub 2004 Mar 17. PMID 15029473
- [Result] Randolph AG, Meert KL, O'Neil ME, Hanson JH, Luckett PM, Arnold JH, Gedeit RG, Cox PN, Roberts JS, Venkataraman ST, Forbes PW, Cheifetz IM; Pediatric Acute Lung Injury and Sepsis Investigators Network. The feasibility of conducting clinical trials in infants and children with acute respiratory failure. Am J Respir Crit Care Med. 2003 May 15;167(10):1334-40. doi: 10.1164/rccm.200210-1175OC. Epub 2003 Feb 25. PMID 12615617
- [Result] Henderson WR, Chen L, Amato MBP, Brochard LJ. Fifty Years of Research in ARDS. Respiratory Mechanics in Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2017 Oct 1;196(7):822-833. doi: 10.1164/rccm.201612-2495CI. PMID 28306327
- [Result] Neto AS, Simonis FD, Barbas CS, Biehl M, Determann RM, Elmer J, Friedman G, Gajic O, Goldstein JN, Linko R, Pinheiro de Oliveira R, Sundar S, Talmor D, Wolthuis EK, Gama de Abreu M, Pelosi P, Schultz MJ; PROtective Ventilation Network Investigators. Lung-Protective Ventilation With Low Tidal Volumes and the Occurrence of Pulmonary Complications in Patients Without Acute Respiratory Distress Syndrome: A Systematic Review and Individual Patient Data Analysis. Crit Care Med. 2015 Oct;43(10):2155-63. doi: 10.1097/CCM.0000000000001189. PMID 26181219
- [Result] Erickson S, Schibler A, Numa A, Nuthall G, Yung M, Pascoe E, Wilkins B; Paediatric Study Group; Australian and New Zealand Intensive Care Society. Acute lung injury in pediatric intensive care in Australia and New Zealand: a prospective, multicenter, observational study. Pediatr Crit Care Med. 2007 Jul;8(4):317-23. doi: 10.1097/01.PCC.0000269408.64179.FF. PMID 17545931
- [Result] Zhu YF, Xu F, Lu XL, Wang Y, Chen JL, Chao JX, Zhou XW, Zhang JH, Huang YZ, Yu WL, Xie MH, Yan CY, Lu ZJ, Sun B; Chinese Collaborative Study Group for Pediatric Hypoxemic Respiratory Failure. Mortality and morbidity of acute hypoxemic respiratory failure and acute respiratory distress syndrome in infants and young children. Chin Med J (Engl). 2012 Jul;125(13):2265-71. PMID 22882846
- [Result] Bellani G, Laffey JG, Pham T, Fan E, Brochard L, Esteban A, Gattinoni L, van Haren F, Larsson A, McAuley DF, Ranieri M, Rubenfeld G, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators; ESICM Trials Group. Epidemiology, Patterns of Care, and Mortality for Patients With Acute Respiratory Distress Syndrome in Intensive Care Units in 50 Countries. JAMA. 2016 Feb 23;315(8):788-800. doi: 10.1001/jama.2016.0291. PMID 26903337
- [Result] Laffey JG, Bellani G, Pham T, Fan E, Madotto F, Bajwa EK, Brochard L, Clarkson K, Esteban A, Gattinoni L, van Haren F, Heunks LM, Kurahashi K, Laake JH, Larsson A, McAuley DF, McNamee L, Nin N, Qiu H, Ranieri M, Rubenfeld GD, Thompson BT, Wrigge H, Slutsky AS, Pesenti A; LUNG SAFE Investigators and the ESICM Trials Group. Potentially modifiable factors contributing to outcome from acute respiratory distress syndrome: the LUNG SAFE study. Intensive Care Med. 2016 Dec;42(12):1865-1876. doi: 10.1007/s00134-016-4571-5. Epub 2016 Oct 18. PMID 27757516